CLINICAL TRIAL: NCT02379403
Title: Effects of Tart Cherry and Aroniaberry Supplementation on Endothelial Function and Cardiovascular Measures in Healthy Older Adults:Interactions With Genotype and Proteome
Brief Title: Effects of Tart Cherry and Aroniaberry Supplementation on Endothelial Function and Cardiovascular Measures in Healthy Older Adults: Interactions With Genotype and Proteome
Status: Withdrawn | Type: Observational
Sponsor: National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 150085; 15-NR-0085
Record Dates: First submitted 2015-03-04; First posted 2015-03-05 (Estimated); Last update posted 2017-10-06 (Actual); Status verified 2017-05-09

CONDITIONS: Cardiovascular Disease; Coronary Heart Disease; Aging
Keywords: Flavonoid; Vascular; Biomarkers; Arterial Stiffness; Nutrigenomics
MeSH Terms: conditions — Cardiovascular Diseases; Coronary Disease

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective

SUMMARY:
Background:

- Heart disease is the leading cause of death and disabilities in the United States. Diets high in fruits and vegetables may reduce the risk of heart disease. Fruits, including red tart cherries and purple aroniaberries, may be especially beneficial. Researchers want to know how tart cherry and aroniaberry extracts affect heart health.

Objective:

- To study the benefits of tart cherry and aroniaberry extract on vascular function and other measures. These include inflammation, oxidation, and cholesterol.

Eligibility:

- Men and post-menopausal women ages 55 70 in good health and with normal or slightly high blood pressure or cholesterol.

Design:

* Participants will be screened with a physical exam, medical history, and blood tests.
* Participants will have 6 visits. They will have blood taken at every visit.
* Visit 1:
* Blood vessel tests. Participants will lie down. Heart rhythm will be monitored. A device will be placed on the upper arm, and pictures of blood vessels will be taken.
* A blood pressure cuff will be tightened around the lower arm for 5 minutes.
* Cardio-Ankle-Vascular Index (CAVI). Blood pressure cuffs will be placed on both arms and legs. They will be tightened with air at the same time for a few minutes.
* Participants will be assigned to one of three groups. For 3 weeks each, in random order, they will take: aroniaberry capsules, tart cherry capsules, placebo capsules, and no capsules.
* Participants will answer questions online about their eating and exercise.
* Participants will be keep a record of what they eat for a few periods. They will come for a study visit every 3 weeks through week 15.

DETAILED DESCRIPTION:
Cardiovascular disease (CVD) continues to be the leading cause of death and disability worldwide. Cardiovascular disease can be age-related in both onset and progression. The aging process causes failure in protective vascular mechanisms leading to pathophysiological changes and increased risk of CVD. Heart healthy strategies including consumption of diets rich in fruits and vegetables reduce risk and prevent CVD. There is growing experimental evidence that certain fruits and berries including, cherries and aroniaberries, may be cardioprotective due to their antioxidant and vasodilatory properties, and beneficial modulation of immune function and inflammation. However, there are limited human studies that have examined these effects. In older adults, vascular aging predominantly includes increased arterial stiffness and endothelial dysfunction. Oxidative stress and inflammation are also linked to the aging process. Therefore, this study will investigate the effects of tart cherry and aroniaberry supplementation on endothelial function (flow-mediated brachial artery dilation) and arterial stiffness (cardio-ankle vascular index) as indicators of cardiovascular risk and atherosclerosis. These measurements also provide an assessment of arterial structure and function. Biomarkers of endothelial dysfunction, inflammation, vascular injury, oxidation, lipids, as well as flavonoid and phenolic acid profiles will also be examined. Importantly, the role of genetics and its environmental interactions as causal factors in CVD are not completely understood. There is also limited data on the plasma proteome and the changes in physiological processes that may result from interventions with diet or nutrients. This study will explore the association between responses to tart cherry or aroniaberry supplementation and single nucleotide polymorphisms (SNPs) in loci related to the study s outcomes and to the risk of CVD. Moreover, the association between these two supplements and a proteomic panel of plasma proteins involved in several physiological pathways and CVD will also be investigated. In a randomized, double-blind, placebo-controlled, crossover clinical trial, 96 healthy older adults (ages 55-70) will be given tart cherry alternating with aroniaberry supplementation daily for 3 weeks each while on their usual diet. This study will include an initial screening visit followed by 6 visits at 3 week intervals consisting of treatment, washout and placebo periods. This investigation will provide important information on the role of flavonoidrich nutrients and their effect on arterial structure and function. Relating genomic and proteomic signatures to the outcomes of this study will be useful in developing future therapeutic strategies to lower CVD risk.

ELIGIBILITY:
* INCLUSION CRITERIA:

An Associate Investigator will examine participants and determine their eligibility according to the inclusion and exclusion criteria as documented by the eligibility checklist.

* Men and women between the ages 55-70 years
* In good general health as determined by physical exam and normal ranges obtained during screening
* Post-menopausal women (no menses within 12 months)
* Normal or pre-hypertensive blood pressure (e.g., SBP less than or equal to 139 mmHg and DBP less than or equal to 89 mmHg)
* Normal or mild hyperlipidemia (e.g., TC less than or equal to 239, LDL less than or equal to159, Triglycerides less than or equal to 199, HDL <45 mg/dL)
* BMI between 18.5 to 25kg/m2
* Willing and ability to sign consent
* Willing to make time commitment for study
* Individuals who are fluent in English

EXCLUSION CRITERIA:

* Progressive or unstable known disease of any body system including cardiovascular, pulmonary, gastrointestinal, central nervous system, psychiatric, endocrine, hematologic, renal, or immunologic disorders
* Known acute and chronic inflammatory disease (i.e. rheumatoid arthritis, systemic lupus erythematous, hepatitis)
* Elevated C-reactive protein level (>3.0mg/L)
* Current (or within the last 3 months) smoking of any tobacco products, i.e., cigarettes, pipe
* Abnormal Complete Metabolic Panel (CMP), Complete Blood Count (CBC), cholesterol panel, Thyroid Stimulating Hormone (TSH), Erythrocyte Sedimentation Rate (ESR) -- (laboratory values outside of acceptable reference range for older adults if determined to

be clinically significant)

* Indications of current or within last 3 years substance or alcohol abuse
* Alcohol consumption >1 drink/day, i.e., 1 bottle of beer, half glass of wine, 1 shot hard liquor
* Known sensitivity or allergy to tart cherry or aroniaberry
* Currently on cholesterol-lowering, anti-hypertensive, thyroid, steroid or hormonal medications
* Routine use of vitamins, supplements, or over the counter medications including aspirin, aspirin-containing products, non-steroidal anti-inflammatory drugs (NSAIDs), i.e., motrin, advil, aleve, unless they were discontinued 14 days prior to their first visit.

Ages: 55 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-02-19; Primary Completion 2017-05-09 (Actual); Study Completion 2017-05-09 (Actual)

PRIMARY OUTCOMES:
Endothelial Function | Every 3 weeks over 15 weeks

SECONDARY OUTCOMES:
Arterial stiffness, biomarkers of endothelial dysfunction, inflammation, vascular injury, oxidation, lipids, nitric oxide status, flavonoid and phenolic acid profiles. | Every 3 weeks over 15 weeks
Proteomic panel of plasma proteins | Every 3 weeks over 15 weeks
Nutrigenomics | Every 3 weeks over 15 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Mary B Engler, Ph.D., Principal Investigator — National Institute of Nursing Research (NINR)

REFERENCES:
- [Background] Engler MB, Engler MM, Chen CY, Malloy MJ, Browne A, Chiu EY, Kwak HK, Milbury P, Paul SM, Blumberg J, Mietus-Snyder ML. Flavonoid-rich dark chocolate improves endothelial function and increases plasma epicatechin concentrations in healthy adults. J Am Coll Nutr. 2004 Jun;23(3):197-204. doi: 10.1080/07315724.2004.10719361. PMID 15190043
- [Background] Tresserra-Rimbau A, Rimm EB, Medina-Remon A, Martinez-Gonzalez MA, de la Torre R, Corella D, Salas-Salvado J, Gomez-Gracia E, Lapetra J, Aros F, Fiol M, Ros E, Serra-Majem L, Pinto X, Saez GT, Basora J, Sorli JV, Martinez JA, Vinyoles E, Ruiz-Gutierrez V, Estruch R, Lamuela-Raventos RM; PREDIMED Study Investigators. Inverse association between habitual polyphenol intake and incidence of cardiovascular events in the PREDIMED study. Nutr Metab Cardiovasc Dis. 2014 Jun;24(6):639-47. doi: 10.1016/j.numecd.2013.12.014. Epub 2014 Jan 22. PMID 24552647
- [Background] Ungvari Z, Kaley G, de Cabo R, Sonntag WE, Csiszar A. Mechanisms of vascular aging: new perspectives. J Gerontol A Biol Sci Med Sci. 2010 Oct;65(10):1028-41. doi: 10.1093/gerona/glq113. Epub 2010 Jun 24. PMID 20576649